CLINICAL TRIAL: NCT07378072
Title: Efficacy of 12-week Daytime Restricted Eating on Hepatic Steatosis of Obesity: Randomized, Open-label, Parallel Group, Controlled Superiority Trial _ CHRONOSTEATOSIS
Brief Title: Efficacy of 12-week Daytime Restricted Eating on Hepatic Steatosis of Obesity
Acronym: CHRONOSTEATOSI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC21_0569
Record Dates: First submitted 2025-12-11; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: MASLD (Metabolic Dysfunction-Associated Steatotic Liver Disease)
Keywords: Time-restricted eating; Obesity; MASLD; circadian rhythms
MeSH Terms: conditions — Intermittent Fasting; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (Experimental): Coaching of the patient by a dietetician for reduction of time of daily food intake to a window of 8 hours per day or less and thus increase of daily fasting to at least 16 hours, in addition to usual dietary counselling to achieve a balanced diet (no calorie restriction) and increase physicial activity as recommended (current guidelines).
  Interventions: Behavioral: Time Restricted Eating
- Usual care only (Active Comparator): Only usual care: usual dietary counselling to achieve a balanced diet (no calorie restriction) and increase physicial activity as recommended (current guidelines).
  Interventions: Behavioral: Usual care only

INTERVENTIONS:
Behavioral: Time Restricted Eating — Coaching of the patient by a dietetician for reduction of time of daily food intake to a window of 8 hours per day or less and thus increase of daily fasting to at least 16 hours, in addition to usual dietary counselling to achieve a balanced diet (no calorie restriction) and increase physicial activity as recommended (current guidelines).
  Arms: Time Restricted Eating
Behavioral: Usual care only — Usual care: dietary counselling to achieve a balanced diet (no calorie restriction) and increase physicial activity as recommended (current guidelines).
  Arms: Usual care only

SUMMARY:
The objective of this study is to demonstrate that an < or equal to 8-hour time-restricted eating (i.e., fasting for at least 16 hours every day), not focusing on reducing caloric intake, reduces intra-hepatic fat in patients with obesity and Metabolic dysfunction-Associated Steatotic liver Disease (MASLD).

DETAILED DESCRIPTION:
Obesity is a growing health problem. The increase in obesity is driving the growing prevalence of metabolic dysfunction-associated steatotic liver disease (MASLD, formerly called non-alcoholic fatty liver disease or NAFLD).

Chronobiology has revealed new risk factors for metabolic disease including MASLD. Proof-of-concept studies showed that time-restricted eating (TRE), a dietary intervention that involves longer fasting periods (typically > 12 h per day) without caloric restriction, reprograms metabolism favorably. The state of the art now justifies clinical trials on clinical populations.

The aim of this randomized, parallel group, controlled study is to test the efficacy of Time Restricted Eating (TRE) implemented with dietary coaching and a dedicated mobile application compared to usual care. The primary endpoint is the evolution of liver fat content quantified by Magnetic Resonance Imaging (MRI).

Patients presenting all inclusion criteria without non-inclusion ciriteria will be included and a Magnetic Resonnance Imaging of the liver will be programmed. Randomization will be performed within 3 months post inclusion after MRI results are obtained. Only patients showing Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) > or equal to 8% will be randomized. Other patients will be withdrawn from study before randomization.

After randomization, both groups will benefit from the standard of care for obesity management and metabolic assessment. Both groups will benefit from dietary counselling to achieve a balanced diet (no calorie restriction) and increase physical activity as recommended. This counselling will be performed by weekly phone calls of a centralized dietetician during a period of 12 weeks. Both groups of patients will use a mobile application to daily register time of first food intake and of time of last food intake (through time-stamped photos of first and last feedings). This will allow to know length of the patient's eating period per 24 hours.

Difference between the 2 groups of patients is only that, in the experimental arm (TRE), patients will additionnaly be instructed to reduce time of daily food intake to a window of 8 hours per day or less and thus increase daily fasting to at least 16 hours. This coaching will be performed during the weekly phone calls of a centralized dietetician.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 30.0 and 49.9 kg/m2
* Age between 18 and 65 years (limits included)
* Sedentary (light-intensity physical activity less than 1 hour per week) or moderately active (moderate exercise 1 to 2 hours per week). Self-declared criteria.
* Weight stable for at least 3 months prior to the beginning of the study (gain or loss <4 kg). Self-declared criteria.
* Able to give written informed consent
* Self-reported eating interval > 12 hours per day
* Subject who owns a smartphone with access to the internet, and agrees to use it in the study
* Affiliation with French social security system or beneficiary from such system
* Fibroscan® Controlled Attenuation Parameter (CAP) > 300 dB/ms
* Hepatitis B and C serologies negative (or showing past-infection or protective immunization)

Exclusion Criteria:

* Alcohol intake > 20 g/day
* Night-shift workers or rotating shift workers
* Smoking
* Patient with diabetes if HbA1c not at target (<7%) and/or using a non-authorized medication)
* Chronic liver disease other than MASLD
* Severe hepatic disease (cirrhosis, hepatocellular carcinoma)
* Severe cardiac disease (Chronic heart failure classified as being in New York Heart Association (NYHA) Class III or IV)
* Severe Kidney disease with CKD-EPI<30 mL/min/1,73m2
* Initiation of hormonal treatment during the study period
* Medications affecting weight or energy balance
* Magnetic Resonance Imaging (MRI) not possible due to patient's anthropometric characteristics. Any of the following:

  * abdominal and/or thoracic circumference with arms greater than 200 cm
  * Sagittal diameter (or abdominal height, i.e. the distance between the dorsum and the apex of the abdomen, which was measured in the supine position at the midpoint between the iliac crest and the last rib) over 70 cm
  * body weight over 160 kg
* MRI not possible due to the following (an MRI safety screening form will have to be filled for inclusion): presence of a pacemaker or cardiac defibrillator or cardiovascular catheter or neurostimulator or an implantable electronic pump for automated drug injection or an electronically-controlled implantable chamber. Ocular metallic foreign bodies
* History of severe eating disorders: Binge Eating Disorder, Bulimia Nervosa; Night eating syndrome
* Minors
* Adults under guardianship, trusteeship or under safeguard of justice
* Other clinical trial participation that could interfere with the study
* Pregnant women or women trying to be pregnant
* Nursing mothers
* Any treatment triggering hepatic steatosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Liver fat content quantified by Magnetic Resonance Imaging Proton Density Fat Fraction | 12 weeks post randomization
  Liver fat content quantified Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) before randomization and then at 12 weeks post randomization

SECONDARY OUTCOMES:
Average lenght of the eating period per 24 hours | 12 weeks post randomization
  Average lenght of the eating period per 24 hours as assessed byt he self-declared times of first and last food intake every day of the 12 weeks intervention. (Daily registration of time of first food intake and of time of last food intake will be performed by all patients on the dedicated mobile application through time-stamped photos of first and last feedings)
Liver steatosis and Stiffness as assessed by the Fibroscan | 12 weeks post randomization
  Liver steatosis ans stiffness evaluated by Fibroscan Controlled Attenuation Parameter before randomization and then at 12 weeks post randomization
Hepatic outcomes evaluated through aspartates aminotransferases (ASAT) blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of aspartate aminotransferases (ASAT) in blood before randomization and at 12 weeks post randomization.
Physical activity level measured by accelerometry with a watch accelerometer | 12 weeks post randomization
  Physical activity measured by accelerometry with a watch accelerometer during 7 days before randomization, then during 7 days of the sixth and twelfth weeks after randomization.
Anthropometric outcomes assessed by body weight. | 12 weeks post randomization
  Patient weight assessed before randomization, then at 6 and 12 weeks post randomization
Anthropometric outcomes assessed by impedancemetry | 12 weeks pour randomization
  Anthropometric oucome : body fat assessed by impedancemetry before randomization, then at 6 and 12 weeks post randomization
Anthropometric outcomes assessed by Magnetic Resonance Imaging of the liver | 12 weeks post randomization
  Percentage of visceral and sub-cutaneaous fat, percentage of muscle fat and muscular surface assessed by Magnetic Resonance Imaging before randomization and at 12 weeks post randomization.
Blood pressure | 12 weeks post randomization
  Blood pressure measured before randomization, then at 6 and 12 weeks post randomization
Metabolic outcomes related to energy balance evaluated through glycated hemoglobin (HbA1c) blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of HbA1c in blood before randomization and at 12 weeks post randomization.
Metabolic outcomes related to energy balance or insulin signaling/resistance assessed through indirect calorimetry | 12 weeks post randomization
  Metabolic outcome : resting energy expenditure as assessed by indirect calorimetry at assessed by indirect calorimetry before randomization then at 12 weeks post randomization.
Depression assessed using the PHQ-9 questionnaire | 12 weeks post randomization
  Depression assessed using the PHQ-9 (Patient Health Questionnaire-9) before randomization , then at 12 weeks post randomization
Anxiety assessed using the GAD-7 questionnaire | 12 weeks post randomization
  Anxiety assessed using the Generalized Anxiety Disorder questionnaire (GAD-7) before randomization, then at 12 weeks post randomization
Quality of sleep using Pittsburgh sleep quality index | 12 weeks post randomization
  Quality of sleep using Pittsburgh sleep quality index before randomization, then at 12 weeks post randomization
Quality of life assessed by EQ-5D questionnaire | 12 weeks post randomization
  Quality of life assessed by the Euro Quality of Life-5 Dimensions (EQ-5D) questionnaire before randomization, then at 12 weeks post randomization.
Chronotype as assessed by Micro Munich ChronoType Questionnaire | 12 weeks post randomization
  Chronotype as assessed by Micro Munich ChronoType Questionnaire before randomization, then at 12 weeks post randomization
Appetite as assessed by FCQ-T-r questionnaire | 12 weeks post randomization
  Appetite as assessed by Food Craving Questionnaire-Trait-reduced (FCQ-T-r) before randomization, then at 12 weeks post randomization
Caloric intake | 12 weeks post randomization
  Total caloric intake and macronutrient repartition as assessed by registration on the dedicated mobile application of photos of patient's intakes during 3 days before randomization, then during 3 days of the sixth and twelfth weeks after randomization
Occurrence of the following adverse events: headache, nausea, diarrhea, constipation, dizziness, fatigue and irritability | 12 weeks post randomization
  Occurrence of the following adverse events: headache, nausea, diarrhea, constipation, dizziness, fatigue and irritability up to 12 weeks post randomization
Hepatic outcomes evaluated through alanine aminotransferase (ALAT) blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of alanine aminotransferase (ALAT) in blood before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through gamma glutamyl-transpeptidase (gamma-GT) blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of gamma glutamyl-transpeptidase (gamma-GT) in blood before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through alcaline phosphatases (ALP) blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of alcaline phosphatases (ALP) in blood before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through bilirubin blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of bilirubin in blood before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through blood parameter transferrin saturation coefficient before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of transferrin saturation coefficient before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through ferritin blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of ferritin in blood before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through blood parameter prothrombin ratio before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of prothrombin ratio before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through iron blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of iron in blood before randomization and at 12 weeks post randomization.
Hepatic outcomes evaluated through protein C-reactive (CRP) blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of protein C-reactive (CRP) in blood before randomization and at 12 weeks post randomization.
Anthropometric outcomes assessed by waist circumference. | 12 weeks post randomization
  Patient waist circumference assessed before randomization, then at 6 and 12 weeks post randomization.
Anthropometric outcomes assessed by hip circumference. | 12 weeks post randomization
  Patient hip circumference assessed before randomization, then at 6 and 12 weeks post randomization.
Metabolic outcomes related to energy balance evaluated through total cholesterol blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of total cholesterol in blood before randomization and at 12 weeks post randomization.
Metabolic outcomes related to energy balance evaluated through LDL-cholesterol blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of LDL-cholesterol in blood before randomization and at 12 weeks post randomization.
Metabolic outcomes related to energy balance evaluated through HDL-cholesterol blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of HDL-cholesterol in blood lbefore randomization and at 12 weeks post randomization.
Metabolic outcomes related to energy balance evaluated through triglycerids blood level before randomization and at 12 weeks post randomization. | 12 weeks post randomization
  Level of triglycerids in blood before randomization and at 12 weeks post randomization.
Metabolic outcomes related to energy balance or insulin signaling/resistance assessed through glucose continuous monitoring | 12 weeks post randomization
  Continous monitroing of glucose in blood during 7 days before randomization and during 7 days of the sixth and of the twelfth weeks after randomization
Metabolic outcomes related to energy balance or insulin signaling/resistance assessed through determination of HOMA-IR | 12 weeks post randomization
  Homesotasis Model Assessment of Insulin Resistance (HOMA-IR) calculated from basal (fasting) glucose and insulin before randomization then at 12 weeks post randomization
Metabolic outcomes related to energy balance or insulin signaling/resistance assessed through determination of HOMA-beta | 12 weeks post randomization
  Homesotasis Model Assessment for Beta-cell function (HOMA-beta) calculated from basal (fasting) glucose and insulin before randomization then at 12 weeks post randomization

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Dijon-Bourgogne, Dijon
  - CHU Lyon, Lyon
  - CHU Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided